CLINICAL TRIAL: NCT07261202
Title: A Preliminary Study Assessing the Effectiveness of a 26 °C Indoor Temperature Limit on Physiological Responses in Children
Brief Title: Impact of Indoor Overheating on Physiological Strain in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University Research Chair, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HEPRU-2025-10-A
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Heat Stress; Physiological Stress; Cognitive Change
Keywords: Indoor overheating; Indoor temperatures; Heat wave; Thermoregulation; Adolescent; Heat strain; Heat vulnerability; Hyperthermia; Youth; Thermal comfort; Physical activity
MeSH Terms: conditions — Heat Stress Disorders; Hyperthermia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure to indoor temperature upper limit of 26°C (Experimental): Participants exposed daylong (6 hours) to an indoor temperature maintained at 26°C and 45% relative humidity (humidex equivalent of 29).
  Interventions: Other: Simulated exposure to indoor overheating
- Exposure to hot indoor environment of 36°C (Experimental): Participants exposed daylong (6 hours) to an indoor temperature maintained at 36°C and 45% relative humidity (humidex equivalent of 45).
  Interventions: Other: Simulated exposure to indoor overheating

INTERVENTIONS:
Other: Simulated exposure to indoor overheating — Children exposed to a 6-hour simulated heat exposure

SUMMARY:
Communities worldwide are experiencing increasing heat extremes that challenge the limits of human thermoregulation, particularly among vulnerable populations such as children. Compared with adults, children are more susceptible to heat related illness due to less efficient thermoregulatory systems and difficulty recognizing early signs of heat stress. In addition, prolonged heat exposure can adversely affect their mental health, contributing to cognitive decline, heightened anxiety, and irritability. As children spend substantial time in hot environments at school and at home, and as these conditions intensify with climate change, actions to safeguard their health are essential. Yet our understanding of heat exposure effects in children remains incomplete, hindering the development of evidence based strategies to protect them.

To address this gap, the investigators aim to evaluate whether an indoor temperature limit of 26 °C (45 percent relative humidity), the upper threshold recommended to protect older adults, can effectively prevent dangerous increases in physiological strain and declines in cognitive function in children during a simulated daylong heatwave. The preliminary study will assess physiological and cognitive responses in children aged 10 to 15 years during a 6 hour exposure (approximating a typical school day) to two conditions: (1) the recommended indoor temperature upper limit (26 °C) and (2) a high heat condition representative of homes and schools without air conditioning during extreme heat events (36 °C). In both conditions, children will remain seated at rest while wearing light clothing (t shirt and shorts), with the exception of performing 15 minutes of stepping exercise (6-6.5 METS) each hour (excluding the lunch period) to reflect typical daily activity in a school setting. This experimental design will allow investigators to determine whether maintaining indoor temperatures at the recommended upper limit for older adults sufficiently mitigates physiological strain in children.

ELIGIBILITY:
Inclusion Criteria:

* English or French speaking.
* Ability to provide informed assent.

Exclusion Criteria:

* Chronic health conditions
* Endurance exercise training (greater than 3 sessions of vigorous exercise training per week for 30 minutes or more)
* Restrictions to physical activity

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-11-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Core temperature (Peak) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Peak rectal temperature (15 min average) during exposure. Rectal temperature is measured continuously throughout the 6 hour exposure to the simulated indoor overheating.
Core temperature (AUC) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Areas under the curve (AUC) of rectal temperature during the 6 hour exposure to the simulate indoor overheating.
Core temperature end of daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Rectal temperature measured at hour 6 of exposure to indoor overheating (15-min average).
Mean skin temperature (Peak) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Peak mean skin temperature (15 min average) during exposure. Mean skin temperature as calculated from skin temperature measured across 7 body regions is measured continuously throughout the 6 hour exposure to the simulated indoor overheating.
Mean skin temperature (AUC) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Areas under the curve (AUC) of mean skin temperature as calculated over 7 body regions during the 6 hour exposure to the simulate indoor overheating.
Mean skin temperature end of daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Mean skin temperature measured over 7 body regions at hour 6 of exposure to indoor overheating (15-min average).
Heat rate (Peak) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Peak heart rate (15 min average) during exposure. Heart rate is measured continuously throughout the 6 hour exposure to the simulated indoor overheating.
Heart rate (AUC) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Areas under the curve (AUC) of heart rate during the 6 hour exposure to the simulate indoor overheating.
Heart rate end of daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Heart rate measured at hour 6 of exposure to indoor overheating (15-min average).
Systolic blood pressure during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Systolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures).
Diastolic blood pressure during daylong exposure to indoor overheating. | At the start (hour 0) and end of 6 hour daylong exposure
  Diastolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures).
Reaction time during daylong exposure to indoor overheating (cognitive function). | At the start (hour 0) and end of 6 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of reaction time. Participants will be asked to initiate a movement of the device in response to a visual cue.
Impulse control during daylong exposure to indoor overheating (cognitive function). | At the start (hour 0) and end of 6 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of impulse control. Participants will be asked to respond to both "go" and "no-go" visual cues. In response to the "go" cue, participants will initiate a movement of the device.
Memory recall during daylong exposure to indoor overheating (cognitive function). | At the start (hour 0) and end of 6 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of memory recall. Participants complete both a delayed recall test and a working memory test.
CDC 4-Stage Balance Test during daylong exposure to indoor overheating (postural stability). | At the start (hour 0) and end of 6 hour daylong exposure
  To assess postural stability, participants hold a tablet to their chest, then auditory cues guide participants through four consecutive stances, feet side by side, instep of one foot touching the big toe of the other foot, tandem stand with one foot in front of the other, heel touching toe, and stand on one foot. The balance assessment will be evaluated based on movement detected by an accelerometer integrated into the hardware of the tablet device (Sway Medical Inc).
Executive function during daylong exposure to indoor overheating (cognitive function). | At the start (hour 0) and end of 6 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of executive function. Participants will complete the Cued Stroop test, in which they are presented a sequence of congruent, neutral and incongruent color-word tasks.
BTrackS Balance Assessment during daylong exposure to indoor overheating (postural stability). | At the start (hour 0) and end of 6 hour daylong exposure
  To assess postural stability, participants will be asked to stand on a BTracks force plate with their feet spread out to shoulder width, hand on their hips and eyes closed. The assessment will comprise of four trials (one practice trial) lasting 20 seconds in length and 20 seconds between trials. Center of pressure (COP) vector data along vertical (y) and horizontal (x) axes will be summed for the total path excursion length (cm) during each trial
Hydration status during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Hydration status measured via assessing the urine specific gravity of a urine sample.
Fluid consumption during daylong exposure to indoor overheating | At end of 6 hour daylong exposure
  Average hourly fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure (normalized to the exposure duration).
Fluid loss during daylong exposure to indoor overheating | At end of 6 hour daylong exposure
  Fluid loss calculated as the change in body mass during each exposure presented as a percentage of baseline body mass (corrected for food consumption).
Thermal sensation scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Thermal sensation assessed via a visual analog scale (How hot do you feel?) ranging from "extremely hot" to "neutral".
Thermal sensation 2 scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Thermal sensation assessed via a visual analog scale ("How do you feel?") ranging from "hot" to "cold"(midpoint: neutral)
Thermal comfort scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") ranging from "very uncomfortable" to "comfortable".
Thirst sensation scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Thirst sensation assessed via a visual analog scale ranging from very, very thirsty to not thirsty at all.
Feel good scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Feel good scale assessed via a visual analog scale (How good do you feel?) ranging from "very good" to "very bad" (midpoint: neutral)
Activity levels during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Activity levels assessed via a wearable monitor (Actical) containing an accelerometer worn on the wrist and hip.
Perceived exertion scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 6 hour daylong exposure
  Perceived exertional assessed via a visual analog scale ("How hard are you working?") ranging from "no exertional at all" to "maximal exertion"

SECONDARY OUTCOMES:
Profiles of Mood States (POMS) during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Potential changes in mood (7 subscales of mood: tension, anger, depression, fatigue, confusion, vigor and esteem related affect). The POMS-40 is a validated, self-administered questionnaire that examines seven distinct aspects of mood state across two positive subscales (Esteem-Related Affect, and Vigor) and five negative subscales (Fatigue, Tension, Confusion, Anger, and Depression), which are described across 40 distinct adjectives. For each individual item, participants were asked to describe "how you feel right now" by responding using a 5-point Likert scale (0 = "Not at all", 1 = "A little", 2 = "Moderately", 3 = "Quite a lot", or 4 = "Extremely"). The values of items associated with a specific subscale (e.g., Fatigue) were summed to calculate its score.
Environmental Symptoms Questionnaire (ESQ) during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Self-reported environmental reactions and medical symptomatology associated with prolonged heat exposure. The ESQ-IV is a validated 68-item, self-administered questionnaire that has been used successfully in identifying symptomatology during exposure to a wide variety of environmental conditions, including heat exposure.
  Participants are asked to assess and described "how you have been feeling today" by responding to each item using a 6-point Likert scale (0 = "Not at all", 1 = "Slight", 2 = "Somewhat", 3 = "Moderate", 4 = "Quite a bit", or 5 = "Extreme"). Total Symptom Score was calculated from this data by taking the sum of the intensity ratings from all 68 individual items using reverse scores for the three positive items from the list ("I Felt Good", "I Felt Alert", and "I Felt Wide Awake").

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada